CLINICAL TRIAL: NCT06066775
Title: A Prospective Cohort Study on the Associations of Endocrine Glucose & Lipids With Brain Aging-related Conditions in Chinese Men and Women
Brief Title: Endocrine Glucose & Lipids Metabolism and Brain Aging: a Longitudinal Study
Status: Recruiting | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Principal Investigator, Shandong Provincial Hospital
Other Study IDs: 20230907
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Brain Aging Related Conditions
Keywords: brain aging; cognition; lipid; glucose
MeSH Terms: interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples were collected and retained for biomarker analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation study without intervention — Observation study without intervention

SUMMARY:
With aging, brain aging leads to a general decline in cognitive ability, and the prevalence of neurodegenerative diseases such as Alzheimer's disease (AD) and Parkinson's disease (PD) increases. The prevalence of abnormal glucose and lipid metabolism also increased with age. The imbalance of glucose and lipid metabolism is closely related to brain aging related conditions and diseases, and the relationship between glucose and lipid metabolism and brain aging has not been fully elucidated.

Phase 1: Baseline investigation (community-based survey) Aims: To investigate whether glucose and lipids are the risk factors for brain aging-related conditions, such as mild cognitive impairment.

Subjects and Methods: A community-based survey will be carried out in 10000 natural population aged >=50 years selected from 10-12 communities stratified according to geographic regions (Ciyao, Huafeng, Dongzhuang, Heshan, Geshi, Jiangji, Gangcheng, Fushan, Dongshu, Sidian, Baxianqiao, and Xiangyin, etc) in Ningyang County, Taian City, Shandong Province. A comprehensive examination including questionnaire (including the MMSE and ADL evaluation for the participants), anthropometric measurements, biochemical analysis will be performed in each study participant. In particular, the investigators randomly selected 1000-2000 participants performing MRI of the brain to evaluate the brain aging related conditions.

Phase 2: Cohort follow-up Aims : To examine glucose and lipids metabolism levels and their changes that modify the risk of brain aging-related conditions.

Subjects and Methods: To recruit and follow all 10000 participants for at least 3-5 years. In particular, all 1000-2000 participants with the baseline MRI examination will perform the MRI examination again for the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 50 years old;
2. Gender: males and females;
3. Provide written informed consent;
4. Satisfactory compliance.

Exclusion Criteria:

1. Pregnant or lactating women
2. No history of addiction or neurological, psychiatric, or systemic diseases known to affect cognitive function, including head trauma, subdural hematoma, current depression, and epilepsy
3. Any other condition or major systemic diseases that the investigator feels would interfere with trial participation or evaluation of results.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In phase 1, 10000 individuals selected from 10-12 communities stratified according to geographic regions. Among them, 1000-2000 individuals receive the MRI examination.
  In Phase 2, 10000 individuals recruited in phase 2 follow-up. Among them, 1000-2000 individuals with the baseline MRI examination will again receive the MRI examination during the follow-up
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
number of participants who develop brain aging-related conditions during follow-up | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Study Chair — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided